CLINICAL TRIAL: NCT00251446
Title: A Phase II Single Arm Trial of Single-agent Vinflunine as Second-line Treatment of Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veeda Oncology (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-05-009
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vinflunine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vinflunine — 320 mg/m2 as a 20-minute IV infusion

SUMMARY:
This is a Phase II, single-arm study in patients with stage IIIB (with malignant pleural effusion) and IV NSCLC who have been previously treated with a platinum-based doublet.

Each cycle will be 21 days. On Day 1 of each cycle, patients will receive vinflunine 320 mg/m2 as a 20-minute IV infusion.

Patients will continue to receive study treatment until disease progression or unacceptable toxicity.

Patients will be evaluated every 2 cycles for response using RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients must fulfill all of the following criteria:

* Patients must have signed an IRB-approved informed consent.
* Patients must have recurrent or metastatic stage IIIB (with malignant pleural effusion) and IV NSCLC that has progressed after receiving a platinum-based doublet as first-line therapy.
* Patients must have measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Previously irradiated lesions will not be allowed as measurable disease.
* Patients must have an ECOG Performance Status of 0, 1, or 2.
* Patients must be <18 years of age.
* Previous chemotherapy must have been completed at least 4 weeks prior to enrollment.
* Patients must either be not of child bearing potential or have a negative serum pregnancy test within 7 days prior to registration. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal for at least 12 months.
* Patients of childbearing potential must agree to use effective contraceptive measures during study treatment and for a reasonable time thereafter.
* Patients must have an absolute neutrophil count (ANC) >1500/uL, platelet count >100,000/uL, and hemoglobin >8 g/dL.
* Patients must have a serum creatinine <2 x institutional upper limit of normal (ULN).
* Patients must have a total bilirubin <2.5 x ULN and aspartate transaminase (AST) <5.0 x ULN.

Exclusion Criteria:

Any of the following criteria will make the patient ineligible to participate in this study:

* Patients previously treated with vinflunine or another vinca alkaloid.
* Patients with untreated and clinically unstable brain metastases.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Patients with a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection.
* Patient has a co-existing malignancy or had a malignancy diagnosed within the last 3 years, with the exception of basal cell carcinoma or cervical cancer in situ.
* Patient received treatment with a non-approved or investigational drug within 30 days before planned start of study treatment.
* Patient is not completely healed from a previous oncologic or other major surgery.
* Patient is receiving or planning to receive any concurrent chemotherapy not indicated in the study protocol or an investigational agent during the study period.
* Patients who have a history of hypersensitivity to vinflunine or any of the components in vinflunine or another vinca alkaloid.
* Any patient who is pregnant or lactating.
* Any patient who is unable to comply with requirements of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To determine the 1-year survival rate in patients with stage IIIB-IV NSCLC receiving single-agent vinflunine who were previously treated with a platinum-based doublet. | unk

SECONDARY OUTCOMES:
To assess response rate (RR) of single-agent vinflunine in patients with stage IIIB-IV NSCLC who were previously treated with a platinum-based doublet. | unk
To assess overall survival in patients with stage IIIB-IV NSCLC receiving single-agent vinflunine who were previously treated with a platinum-based doublet. | unk
To determine the progression-free survival (PFS) in patients with stage IIIB-IV NSCLC receiving single-agent vinflunine who were previously treated with a platinum-based doublet | unk
To assess time to response (TTR) in patients with stage IIIB-IV NSCLC receiving single-agent vinflunine who were previously treated with a platinum-based doublet. | unk
To assess duration of overall response in patients with stage IIIB-IV NSCLC receiving single-agent vinflunine who were previously treated with a platinum-based doublet. | unk
To assess duration of stable disease in patients with stage IIIB-IV NSCLC receiving single-agent vinflunine who were previously treated with a platinum-based doublet. | unk
To assess the safety of single-agent vinflunine in patients with stage IIIB-IV NSCLC who were previously treated with a platinum-based doublet. | unk

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Joppert, MD, Principal Investigator — Veeda Oncology
Locations (1):
- Veeda Oncology, Houston, Texas, United States